CLINICAL TRIAL: NCT03053414
Title: A Vitamin D Dosing Strategy for Adequate Repletion and Maintenance in IBD Patients With Minimal Disease Activity
Brief Title: Vitamin D Repletion and Maintenance in IBD: How Much and How Often
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: change in study design before recruitment began
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Eric Vasiliauskas, Associate Clinical Director, Inflammatory Bowel Disease Program, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00045446
Record Dates: First submitted 2017-02-06; First posted 2017-02-15 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Inflammatory Bowel Diseases; Vitamin D Deficiency
MeSH Terms: conditions — Inflammatory Bowel Diseases; Vitamin D Deficiency | interventions — Vitamin D; Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of four treatment arms for the duration of the study. Labs will be checked every 3 months as part of standard of care to help delineate the best strategy for repletion and maintenance of Vitamin D levels throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment Arm # 1 (Active Comparator): 50,000 IU oral vitamin D2 per week for 12 weeks + Dietary counseling
  Interventions: Dietary Supplement: Vitamin D (ergocalciferol and/ or cholecalciferol)
- Treatment Arm # 2 (Active Comparator): 50,000 IU oral vitamin D2 per week x 12 weeks then 800 IU/day oral vitamin D3 for 6 months + Dietary counseling
  Interventions: Dietary Supplement: Vitamin D (ergocalciferol and/ or cholecalciferol)
- Treatment Arm # 3 (Active Comparator): 50,000 IU oral vitamin D2 per week x 12 weeks then 5,000 IU/day oral vitamin D3 for 6 months+ Dietary counseling
  Interventions: Dietary Supplement: Vitamin D (ergocalciferol and/ or cholecalciferol)
- Treatment Arm # 4 (Active Comparator): 5,000 IU oral daily vitamin D3 for 9 months + Dietary counseling
  Interventions: Dietary Supplement: Vitamin D (ergocalciferol and/ or cholecalciferol)

INTERVENTIONS:
Dietary Supplement: Vitamin D (ergocalciferol and/ or cholecalciferol) — To evaluate effective repletion and supplementation for Vitamin D levels in patients with inflammatory bowel disease.

SUMMARY:
Inflammatory bowel disease (IBD), which includes ulcerative colitis (UC) and Crohn's disease (CD), are chronic relapsing inflammatory conditions of the gastrointestinal tract. IBD is thought to result from a complex interaction between genetic, immune, microbial and environmental factors. There is emerging data suggesting Vitamin D may not only play a role in bone health but may also be involved in gut health as well. While there are guidelines regarding the recommending doses of Vitamin D for supplementation and maintenance in bone health, these strategies are unknown in those with inflammatory bowel disease. The investigators seek to determine a dosing strategy for this population using doses within the recommended guidelines for bone health.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD), which includes ulcerative colitis (UC) and Crohn's disease (CD), are chronic relapsing inflammatory conditions of the gastrointestinal tract. IBD is thought to result from a complex interaction between genetic, immune, microbial and environmental factors. The role of vitamin D in bone health and calcium homeostasis is well documented. However, emerging data suggests that vitamin D may also regulate immune responses, which may play a role in the pathogenesis and disease activity of IBD.

The investigators seek to identify CD or UC patients with mild disease or in clinical remission who have vitamin D levels <30 ng/ml and not on any type of vitamin repletion therapy. The investigators will randomize the participants into one of four arms: (1) Oral 50,000 vitamin D IU every week for 12 weeks (2) Oral 50,000 vitamin D weekly for 12 weeks than oral 800 vitamin D IU/d (3) Oral 50,000 vitamin D IU weekly for 12 weeks then 5,000 vitamin D IU/d (4) Oral 5,000 vitamin D IU/d and check vitamin D levels and inflammatory markers as part of standard of care follow- up every 3 months for nine months. Every participant will receive dietary counseling throughout the study duration. Our aim is to identify an optimal dosing strategy for repletion and maintenance of vitamin D levels in the subset of IBD patients. Based on clinical experience, doses higher than the recommended doses for bone health are needed to achieve and maintain optimal levels of Vitamin D in IBD patients, even patients are in remission or do not have small bowel (malabsorption) involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Crohn's disease or Ulcerative colitis
2. In clinical remission or with mild disease activity as determined by the Harvey Bradshaw Index (CD) ≤7 or Ulcerative Colitis disease activity index ≤6.
3. 25(OH)D level <30 ng/ml within three months of study enrollment
4. Provided verbal consent
5. 18 years of age or older

Exclusion Criteria:

1. Unwilling to provide consent or lack capacity
2. Moderate to severe disease activity (Harvey Bradshaw index >7 or UCDAI >6)
3. Current pregnancy or attempting to conceive
4. Known coexisting hyperparathyroidism
5. Already on vitamin D supplementation, calcium supplementation or a multivitamin
6. BMI >30 kg/m²
7. History of kidney stones
8. Subjects <18 years of age - pediatric population with different recommended dosing than adults (10).
9. Non-english speakers

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-20 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Vitamin D levels after completion of repletion dosing | 3 months

SECONDARY OUTCOMES:
Vitamin D levels on maintenance dosing | 9 months

OTHER OUTCOMES:
Medication compliance among participants | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xavier RJ, Podolsky DK. Unravelling the pathogenesis of inflammatory bowel disease. Nature. 2007 Jul 26;448(7152):427-34. doi: 10.1038/nature06005. PMID 17653185
- [Background] Ananthakrishnan AN. Epidemiology and risk factors for IBD. Nat Rev Gastroenterol Hepatol. 2015 Apr;12(4):205-17. doi: 10.1038/nrgastro.2015.34. Epub 2015 Mar 3. PMID 25732745
- [Background] Cantorna MT. Vitamin D, multiple sclerosis and inflammatory bowel disease. Arch Biochem Biophys. 2012 Jul 1;523(1):103-6. doi: 10.1016/j.abb.2011.11.001. Epub 2011 Nov 10. PMID 22085500